CLINICAL TRIAL: NCT06361589
Title: Real World Study of Lolatinib for Patients With Advanced/Metastatic Anaplastic Lymphoma Kinase (ALK) - Positive Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Real World Study of Lolatinib for Advanced ALK+ NSCLC Patients
Status: Recruiting | Type: Observational
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Juan LI, MD, Principal Investigator, Sichuan Cancer Hospital and Research Institute
Other Study IDs: EK2023003-1
Record Dates: First submitted 2024-03-26; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: ALK-positive Non-small Cell Lung Cancer; Real World Study
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Advanced ALK+ NSCLC Patients
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — lolatinib 100mg qd po

SUMMARY:
This study was a multicenter, prospective, non-interventional clinical study that included first-line and late-line patients with advanced non-small cell lung cancer with ALK fusions treated with the third generation ALK-TKI lorlatinib until disease progression, intolerable toxicity, investigator or subject decision to withdraw, lost to follow-up, initiation of other antineoplastic therapy, or death. Clinical pathology including sex, age, ALK mutation status at diagnosis, and clinical stage at diagnosis were collected from medical records. Physical condition as assessed by ECOG-PS before administration of lorlatinib was also recorded. Treatment information was obtained from the records, including dose and timing of ALK-TKI therapy and tumor response, number of prior systemic lines of therapy, and local treatment modalities such as radiotherapy and surgery. Quality of life based on the EORTC QLQ C30+LC29 scale (plus the EORTC QLQ BN20 scale in patients with brain/meningeal metastases) was performed at baseline and at each follow-up point. This study will use REDCap platform to collect and manage the study data information of multi-center patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this clinical study, understanding of study procedures, and ability to sign written informed consent.
2. Age ≥18 years.
3. Locally advanced or metastatic (inoperable stage IIIa or IIIb-IV) NSCLC with disease staging according to the American Joint Committee on Cancer (AJCC)/UICC 8th edition lung cancer staging criteria.ALK fusion mutations confirmed by tumor histology or hematology.
4. Expected survival greater than 12 weeks.
5. Adequate bone marrow reserve, organ function, and coagulation as assessed by the investigator as evidenced by complete blood count, biochemical parameters in blood and urine, coagulation, and electrocardiogram or cardiac ultrasound at baseline.
6. Can take the medicine orally and swallow it.
7. Female patients of childbearing potential are willing to use appropriate contraception and should not breastfeed within 6 months from signing the main informed consent to efficacy evaluation/end of medication (whichever is later); Male patients were willing to use barrier contraception (i.e., condom) for 6 months from signing the main informed consent until the efficacy assessment/end of medication, whichever occurred later.
8. Female patients have a negative blood pregnancy test within 3 days before enrollment or meet one of the following criteria to demonstrate no risk of pregnancy: a. Postmenopausal is defined as age 50 years or older and amenorrhea for at least 12 months after cessation of all exogenous hormone replacement therapy; b. Females less than 50 years of age may also be considered postmenopausal if they have been amenorrhoeic for 12 months or more after cessation of all exogenous hormonal therapy and have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels within the laboratory postmenopausal reference values; c. History of irreversible sterilization, including hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, except for bilateral tubal ligation.

Exclusion Criteria:

1. Use of strong CYP3A4 inhibitors, strong inducers, or drugs with a narrow therapeutic window that are sensitive substrates of CYP3A4 within 7 days and need to continue treatment with these drugs during the study.
2. Patients with known active infectious diseases, such as active hepatitis B or C or HIV infection of human immunodeficiency virus, active hepatitis B and C including hepatitis B or C surface antigen (+) patients receiving intravenous treatment for infection - patients receiving oral antiviral suppression of hepatitis B or C will be allowed to participate in the study.
3. Any other disease, metabolic abnormality, physical examination abnormality, or laboratory abnormality that, in the judgment of the investigator, has reason to suspect that the patient has a disease or condition that is not appropriate for the use of lorlatinib, or would affect the interpretation of the study results, or place the patient at high risk.
4. Female patients who are pregnant, breastfeeding, or plan to become pregnant during the study.
5. Patients with hypersensitivity to any active or inactive ingredient of lorlatinib.
6. Any other patient who, in the judgment of the investigator, may have poor compliance with the study procedures and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients with ALK-mutated non-small cell lung cancer were included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of receiving therapy until date of disease progression or death.Approximately 5 years following the first dose of study drugs
  Intracranial and systemic PFS as assessed by the investigators using RECIST V1.1 or RANO-BM Separately.

SECONDARY OUTCOMES:
OS | From date of receiving therapy until date of death.Approximately 5 years following the first dose of study drugs
  Overall survival for first-line and late-line of lorlatinib medication
ORR | From date of receiving therapy until date of disease progression or the end of study, up to approximately 5 years.
  the Sum of percentage of participants with CR and PR as assessed by RECIST v1.1 or RANO-BM criteria every 8-12 weeks.
AE | Approximately 5 years following the first dose of study drugs.
  Number and percentage of participants with treatment-related AEs as assessed by CTCAE v5.0, and the duration of AEs on every grade.
PRO1 | Approximately 5 years following the first dose of study drugs.
  Change from baseline in quality of life of patients on EORTC QLQ-C30 at every 8-12 Weeks.
PRO2 | Approximately 5 years following the first dose of study drugs.
  Change from baseline in quality of life complemented by EORTC QLQ-LC29 at every 8-12 Weeks.
PRO3 | Approximately 5 years following the first dose of study drugs.
  Change from baseline in activities of daily living of patients with CNS metastases on EORTC QLQ-BM20 at every 8-12 Weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan cancer hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No